CLINICAL TRIAL: NCT07252739
Title: KEYMAKER-U01 Substudy 01J: A Randomized Phase 2 Umbrella Study With Rolling Arms of Investigational Agents for First-line Treatment of Participants With Advanced or Metastatic Nonsquamous Non-small Cell Lung Cancer (NSCLC) With KRAS G12C Mutations
Brief Title: KEYMAKER-U01 Substudy 01J: A Study of Pembrolizumab Plus MK-1084 in Participants With Non-Small Cell Lung Cancer (NSCLC) With Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) G12C Mutations (MK-3475-01J/KEYMAKER-U01J)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3475-01J; U1111-1321-3999 (Registry Identifier: UTN); 2025-521939-36-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2025-11-20; First posted 2025-11-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Malignant Neoplasm
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cetuximab; Carboplatin; Pemetrexed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Some outcome measures will be assessed by blinded independent central review (BICR), with assessor(s) blinded to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Participants receive 400 mg of Pembrolizumab every 6 weeks, Carbo platin every 3 weeks and 500 mg/m^2 of Pemetrexed every 3 weeks.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed
- Arm 2 (Experimental): Participants receive 400 mg of Pembrolizumab every 6 weeks, and MK-1084 dose regimen
  Interventions: Drug: MK-1084; Biological: Pembrolizumab
- Arm 3 (Experimental): Participants receive 400 mg of Pembrolizumab every 6 weeks, 500 mg/m^2 Cetuximab every 2 weeks, and MK-1084 dose regimen
  Interventions: Drug: MK-1084; Biological: Pembrolizumab; Biological: Cetuximab

INTERVENTIONS:
Drug: MK-1084 — Oral Administration
  Arms: Arm 2; Arm 3
Biological: Pembrolizumab — Intravenous administration
  Other Names: Keytruda; MK-3475
Biological: Cetuximab — Intravenous administration
  Arms: Arm 3
Drug: Carboplatin — Intravenous administration
  Arms: Arm 1
Drug: Pemetrexed — Intravenous administration
  Arms: Arm 1

SUMMARY:
Researchers want to learn if using a study medicine called MK-1084 can help treat NSCLC. MK-1084 is a type of treatment called targeted therapy for the Kirsten rat sarcoma viral oncogene homolog (KRAS) G12C gene change. The goal of this study is to learn about the safety of MK-1084 and to learn how many people have the cancer get smaller or go away during the study treatment.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically or cytologically confirmed diagnosis of advanced or metastatic nonsquamous Non-Small Cell Lung Cancer (NSCLC)
* Has tumor tissue or circulating tumor deoxyribonucleic acid (ctDNA) that demonstrates the presence of Kirsten rat sarcoma viral oncogene homolog (KRAS) G12C mutations
* Can provide an archival tumor tissue sample or newly obtained core, incisional, excisional biopsy of a tumor lesion not previously irradiated
* Has recovered to ≤Grade 1 or baseline from any Adverse events (AEs) due to previous anticancer therapies and/or ≤Grade 2 neuropathy and/or endocrine-related AEs adequately treated with hormone replacement
* Has well controlled human immunodeficiency virus (HIV) on antiretroviral therapy (ART) if HIV-infected
* Has undetectable hepatitis B (HBV) viral load and have received HBV antiviral therapy for at least 4 weeks if hepatitis B surface antigen (HBsAg) positive
* Has undetectable hepatitis C (HCV) viral load if HCV-infected

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements
* Has HIV-infection with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous clear history of inflammatory bowel disease
* Has uncontrolled, clinically significant cardiovascular disease or cerebrovascular disease, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, uncontrolled symptomatic arrhythmia, prolongation of corrected QT interval corrected for heart rate by Fridericia's formula (QTcF) interval to >470 ms, and/or other serious cardiovascular and cerebrovascular diseases within the 6 months preceding study intervention
* Has received prior systemic anticancer therapy for advanced or metastatic NSCLC
* Has received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event (irAE) (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis
* Has received previous treatment with an agent targeting KRAS
* Has received prior systemic anticancer therapy within 4 weeks or 5 half-lives (whichever is shorter) and has not recovered to grade ≤ 1 or baseline from AE associated with anticancer therapy before allocation/randomization
* Has received radiation therapy to the lung that is >30 Gray within 6 months of start of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has a known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid) is allowed
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has a history of stem cell/solid organ transplant
* Has not adequately recovered from major surgery or has ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2033-01-14 (Estimated); Study Completion 2033-01-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with a Dose Limiting Toxicity (DLT) | Up to approximately 21 days
  A DLT is defined as the occurrence of protocol-specified toxicities if assessed by the investigator to be possibly, probably, or definitely related to study intervention administration, excluding toxicities clearly not related to the drug.
Percentage of Participants who Experience at Least One Adverse Event (AE) | Up to approximately 84 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Percentage of Participants who Discontinue Study Intervention Due to an AE | Up to approximately 84 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Objective Response Rate (ORR) per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 as assessed by Blinded Independent Central Review (BICR) | Up to approximately 84 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by BICR will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) per RECIST 1.1 as assessed by BICR | Up to approximately 84 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression Free Survival (PFS) per RECIST 1.1 as assessed by BICR | Up to approximately 84 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 84 months
  OS, defined as the time from first dose or randomization (depending on study period) to death due to any cause. OS will be presented.
Area Under the Concentration-Time Curve (AUC) for MK-1084 | At designated timepoints (up to approximately 44 days)
  Blood samples will be collected to determine the AUC of MK-1084.
Maximum Concentration (Cmax) of MK-1084 | At designated timepoints (up to approximately 44 days)
  Blood samples will be collected to estimate Cmax of MK-1084.
Trough Concentration (Ctrough) of MK-1084 | At designated timepoints (up to approximately 84 months)
  Blood samples will be collected to determine the Ctrough of MK-1084.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (9):
- Clermont Oncology Center ( Site 0041), Clermont, Florida, United States
- Severance Hospital Yonsei University Health System ( Site 0080), Seoul, South Korea
- Ukraine (7):
  - COMMUNAL NONPROFIT ENTERPRISE "CLINICAL CENTER OF ONCOLOGY, HEMATOLOGY, TRANSPLANTOLOGY AND PALLIATI ( Site 0139), Cherkasy, Cherkasy Oblast
  - Medical Center "Mriya Med-Service"-Clinical Research Department ( Site 0465), Kryvyi Rih, Dnipropetrovsk Oblast
  - Communal Non-Commercial Enterprise "Prykarpatski Clinical On-Surgery department #2 ( Site 0132), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Limited Liability Company Ukrainian Center of Tomotherapy-Department of Chemotherapy ( Site 0467), Kropyvnytskyi, Kirovohrad Oblast
  - Communal Noncommercial Enterprise "Podillia Regional Oncolog-Cardiothoracic department ( Site 0131), Vinnitsya, Vinnytsia Oblast
  - VISION PARTNER Medical Centre ( Site 0135), Kyiv
  - LIMITED LIABILITY COMPANY "MEDICAL CENTER "DOBROBUT-CLINIC" ( Site 0138), Kyiv

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/